CLINICAL TRIAL: NCT00273611
Title: Characterization of Vitamin D Levels and Affect of Pharmacist-initiated Vitamin D Education in Geriatric Outpatients.
Brief Title: Vitamin D Levels and Vitamin D Education in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 05-0799; 5M01RR000051 (NIH)
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Vitamin D Insufficiency; Vitamin D Deficiency
Keywords: vitamin D deficiency; geriatric patients
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist education (Experimental): Pharmacist education about vitamin D
  Interventions: Behavioral: Pharmacist Education about Vitamin D
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Pharmacist Education about Vitamin D
  Arms: Pharmacist education

SUMMARY:
Vitamin D is important to maintain good health. Although it is found in foods and vitamins, many people still have low vitamin D levels. One purpose of this study is to describe vitamin D levels from patients at the University of Colorado Seniors Clinic. Another goal of the study is to find out if education by a pharmacist can increase vitamin D levels in patients who have low vitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the University of Colorado Hospital Seniors Clinic with an appointment in December 2005 or January 2006
* Age 65-89 years

Exclusion Criteria:

* History of dementia or memory loss
* Severe illness or life expectancy less than 6 months
* Assistance with medications from an assisted living facility
* History of celiac Sprue, Crohn's disease, or chronic pancreatitis
* High calcium levels, high parathyroid hormone levels, low phosphorus levels, or very high vitamin D levels
* Taking prescription vitamin D

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
25(OH) vitamin D level | 12 weeks
  Change in vitamin D level after usual care or pharmacist education

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Linnebur, Pharm.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital Seniors Clinic, Aurora, Colorado, United States

REFERENCES:
- [Result] Vande Griend JP, Linnebur SA, Ruscin JM, Vondracek SF, Wolfe P, McDermott MT. Vitamin D intervention by pharmacists in geriatric outpatients. J Am Pharm Assoc (2003). 2008 Jul-Aug;48(4):501-7. doi: 10.1331/JAPhA.2008.07056. PMID 18653426